CLINICAL TRIAL: NCT03137654
Title: Sex Differences, Cognitive Training & Emotion Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB201700206-N; R03AA025430 (NIH)
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Alcohol Use Disorder
Keywords: Cognitive Training; Emotion Processing
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: The primary design is a 3 (Training Condition: Neutral, Affective, Control) by 2 (Time: Baseline, Post-training) repeated measures design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Affective Training (Active Comparator): Subjects complete baseline assessment, 3 wks of training with versions of the tasks using emotionally-laden stimuli, and a post-training assessment. Subjects will be contacted monthly for 3 months after discharge for follow-up interviews.
  Interventions: Other: Affective Training
- Neutral Training (Active Comparator): Subjects complete baseline assessment, 3 wks of training with versions of the tasks using neutral stimuli, and a post-training assessment. Subjects will be contacted monthly for 3 months after discharge for follow-up interviews.
  Interventions: Other: Neutral Training
- Control (Non-active) (No Intervention): Subjects complete a baseline assessment and a secondary assessment approximately three weeks later. No active intervention is delivered. Subjects will be contacted monthly for 3 months after discharge for follow-up interviews.

INTERVENTIONS:
Other: Affective Training — Intervention includes up to 12 training sessions (~45 minutes each). Training sessions includes practice on cognitive tasks embedded with emotionally salient stimuli. Tasks include a dual modality n-back and a directed attend/ignore memory task.
  Arms: Affective Training
Other: Neutral Training — Intervention includes up to 12 training sessions (~45 minutes each). Training sessions includes practice on cognitive tasks embedded with neutral stimuli. Tasks include a dual modality n-back and a directed attend/ignore memory task.
  Arms: Neutral Training

SUMMARY:
This pilot project addresses two understudied questions related to neurocognitive deficits observed in treatment-seeking alcoholics. First, whether cognitive training improves performance and outcomes in alcoholics, and whether men and women differ in their response to this training. The second is whether directed training using affective materials (e.g., emotional faces) is differentially effective compared to that using traditional (i.e., neutral) stimuli.

DETAILED DESCRIPTION:
This pilot project leverages the team's expertise in neurobehavioral assessment and focus on sex differences to examine the potential efficacy of cognitive training in treatment-seeking men and women with alcohol use disorders (AUDs). Specifically, the ask whether cognitive training interventions derived from current methods and conceptual models has differential benefits for treatment-seeking women vs. men. Although neurocognitive improvement during training is desired, of practical import is whether gains achieved transfer to other tasks and settings. Therefore, transfer of gains to tasks/domains varying in their similarity to training are assessed. Given noted sex differences in emotional processing and the purported role of emotional factors in women's substance use, training engaging emotional processing via the use of affective stimuli (faces and words) is included, predicting that women may differentially benefit from such training. Equal numbers of treatment-seeking men and women with AUDs will be randomly assigned to one of two active training interventions (neutral or affective stimuli). To control for abstinence-related recovery, a third group of participants, meeting identical selection criteria, will complete pre and post-intervention testing, but will not undergo the training intervention. Ss will complete baseline, 3 wks training (for active groups) and post-intervention testing and will be contacted monthly for 3 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 10 years of education
* Subjects must have 20/40 or better corrected vision (determined by Snellen chart)
* have no significant hearing impairment as determined by self-report and audiometric testing
* must meet criteria for DSM-IV alcohol dependence using the computerized Diagnostic Interview Schedule - IV
* A craving index is also administered to allow discussion in terms of DSM 5 classification.
* Comorbid substance use including nicotine use is not exclusionary.

Exclusion Criteria:

* May not have medical or psychiatric histories which would confound participation or data interpretation, e.g., epilepsy, stroke, untreated hypertension, psychotic disorders, anxiolytic medications.
* not be color blind (as determined by psuedoisochromatic plates)
* Endorsement of suicidal intent

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Jo Nixon, PhD, Principal Investigator — University of Florida; Ben Lewis, PhD, Principal Investigator — University of Florida
Locations (5):
- United States (5):
  - ASPIRE Healthcare Facilities, Gainesville, Florida
  - The Sid Martin Bridge House, Gainesville, Florida
  - UF Health Florida Recovery Center, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Steward-Marchman-Act (SMA) Healthcare, Multiple Locations, Florida

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 82 individuals were enrolled in the study. 5 were enrolled, but not started. 77 individuals were started.
Period: Overall Study
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Started | 23 | 25 | 29
Completed | 15 | 13 | 14
Not Completed | 8 | 12 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Affective Training | Neutral Training | Control (Non-active) | Total
Number analyzed (Participants) | 15 | 13 | 14 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.93 (11.70) | 45.62 (12.86) | 39.23 (11.64) | 42.61 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 1 | 9
  Male | 11 | 9 | 13 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 3 | 3 | 1 | 7
  White | 9 | 9 | 11 | 29
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2 | 4
Depressive Symptoms [Mean (Standard Deviation); unit: units on a scale] — Beck Depression Inventory-II
  Total Range = 0-63
  Higher values represent greater depressive symptomatology
  units on a scale | 22.36 (12.01) | 17.18 (9.47) | 20.92 (20.37) | 20.37 (11.33)
Anxiety Symptoms [Mean (Standard Deviation); unit: units on a scale] — Spielberger State Anxiety Index (age-adjusted)
  Total Range = 20-80
  Higher scores indicate greater anxiety symptomatology
  units on a scale | 63.40 (18.06) | 56.83 (16.19) | 68.43 (10.27) | 63.20 (15.56)
Drinks/day [Mean (Standard Deviation); unit: drinks per day] — Standard drinks of alcohol per day (averaged over 6 months)
  drinks per day | 20.84 (19.71) | 16.34 (13.96) | 22.30 (20.49) | 19.94 (18.14)
Maximum Drinks [Mean (Standard Deviation); unit: maximum drinks] — Greatest number of standard drinks consumed within a 24-hour period and occuring within the 6 months prior to treatment initiation
  maximum drinks | 31.75 (19.55) | 26.46 (23.93) | 35.52 (30.04) | 31.26 (24.39)

OUTCOME MEASURES:

1. Primary Outcome: Emotional Stroop: Change From Baseline in Reaction Time
Description: An interference task involving target words presented over non-target visual stimuli. The primary dependent measure is change in reaction time on trials with incongruent stimuli (e.g., a negative word presented over a "happy" face) from baseline to post-training assessment. Change scores are calculated by subtracting reaction time at post-training assessment from reaction time at baseline, thus positive values indicate improvements in processing speed from pre- to post-training (e.g., 500ms [baseline score] - 300ms [post-training score] = 200ms [positive change score]).
Time Frame: Baseline and Post-Training (3 weeks)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Number analyzed (Participants) | 15 | 13 | 14
milliseconds | 336 (378) | 162 (713) | 78.3 (190)
Statistical Analysis 1: Comparison: Affective Training vs Neutral Training vs Control (Non-active); Test type: Superiority; p = .0078, Linear Mixed Model

2. Primary Outcome: Trail-Making Task A: Change From Baseline in Task Completion Time
Description: A psychomotor and visual perception task wherein participants connect numbered dots by drawing a continuous line. The primary dependent measure is change in task completion time from baseline to post--training assessment.
Time Frame: Baseline and Post-Training (3 weeks)
Population: Due to time constraints involved with testing, we removed this tast from the protocol prior to study initiation
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Trail-Making Task B: Change From Baseline in Task Completion Time
Description: A psychomotor and visual perception task with a set-shifting component wherein participants connect numbered and lettered dots by drawing a continuous line. The primary dependent measure is change in task completion time from baseline to post-training assessment.
Time Frame: Baseline and Post-Training (3 weeks)
Population: Due to time constraints involved with testing, we removed this tast from the protocol prior to study initiation
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Digit Symbol Substitution: Change From Baseline in Translated Symbols
Description: A psychomotor and set-shifting task involving translation between numbers and symbols. The primary dependent measure is the change in number of correctly translated symbols within 90 seconds from baseline to post-training assessment.
Time Frame: Baseline and Post-Training (3 weeks)
Population: Due to time constraints involved with testing, we removed this tast from the protocol prior to study initiation
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Number analyzed (Participants) | 0 | 0 | 0

5. Primary Outcome: Little Man Task: Change From Baseline in Response Accuracy.
Description: A visual perception task involving mental rotation. The primary dependent measure is the change in response accuracy from baseline to post-training assessment. This change was calculated as the difference between the proportion of correct responses at baseline and post-training asssessments. Positive values represent gains in accuracy. Negative values represent decreases in accuracy.
Time Frame: Baseline and Post-Training (3 weeks)
Measure: Mean (Standard Deviation); unit: proportion of correct responses
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Number analyzed (Participants) | 7 | 6 | 11
proportion of correct responses | -.0045 (.129) | .125 (.192) | .0483 (.174)
Statistical Analysis 1: Comparison: Affective Training vs Neutral Training vs Control (Non-active); Test type: Superiority; p = 0.393, ANOVA

6. Primary Outcome: Wisconsin Card Sorting Task: Change From Baseline in Response Accuracy
Description: A reasoning and set-shifting task. Participants must determine novel rule sets for stimuli matching through trial and error. Ss must match each 'Test Card' with a 'Key Card'. Criteria for a successful match shift throughout the testing session and may include color, shape, and number of symbols. The primary dependent measure is the change in response accuracy from baseline to post-training assessment.
Time Frame: Baseline and Post-Training (3 weeks)
Population: Data from this task were corrupted, precluding any analysis
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Number analyzed (Participants) | 0 | 0 | 0

7. Primary Outcome: Sternberg Working Memory Task: Change From Baseline in Response Accuracy
Description: A working memory task involving numbers presented visually. Ss are presented with a list of digits, one at a time, followed by a probe digit. They must determine if the probe digit was in the original set of digits and recall the digits. The primary dependent measure is the change in response accuracy (proportion of correct responses) from baseline to post-training assessment. Positive values indicate greater proportions of correct responses at post-test, relative to baseline.
Time Frame: Baseline and Post-Training (3 weeks)
Measure: Mean (Standard Deviation); unit: proportion of correct responses
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Number analyzed (Participants) | 10 | 7 | 9
proportion of correct responses | .0021 (.142) | 0.0298 (.0623) | 0.148 (0.121)
Statistical Analysis 1: Comparison: Affective Training vs Neutral Training vs Control (Non-active); Test type: Superiority; p = .0344, ANOVA

8. Primary Outcome: Stroop Color-Word Task: Change From Baseline in Response Time
Description: An interference task involving target words (e.g., red) presented in interfering colors (e.g., blue). The primary dependent measure is change in reaction time from baseline to post-training assessment. Change scores are calculated by subtracting reaction time at post-training assessment from reaction time at baseline, thus positive values indicate improvements in processing speed from pre- to post-training (e.g., 500ms [baseline score] - 300ms [post-training score] = 200ms [positive change score]).
Time Frame: Baseline and Post-Training (3 weeks)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Number analyzed (Participants) | 7 | 2 | 9
seconds | 5 (25.9) | -11.5 (67.2) | 22 (77.1)
Statistical Analysis 1: Comparison: Affective Training vs Neutral Training vs Control (Non-active); Test type: Superiority; p = .0344, ANOVA

9. Primary Outcome: Visual-Perceptual Analysis Task: Change From Baseline in Response Time
Description: A discrimination task in which participants are asked to determine which complex shape differs among a set of three. Outcomes reflect the difference in response times from baseline to post-test assessments, with negative values corresponding to improved speed at post-test.
Time Frame: Baseline and Post-Training (3 weeks)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Number analyzed (Participants) | 12 | 9 | 8
milliseconds | -1270 (1111) | 121 (1512) | -377 (772)
Statistical Analysis 1: Comparison: Affective Training vs Neutral Training vs Control (Non-active); Test type: Superiority; p = 0.0365, ANOVA

10. Secondary Outcome: Timeline Follow-back
Description: Measures frequency and quantity of daily alcohol use, measured as average ounces of alcohol consumed per day.
Time Frame: 30 days following post-training assessment, up to 1.5 months
Measure: Mean (Standard Deviation); unit: ounces of absolute ethanol per day
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Number analyzed (Participants) | 5 | 5 | 4
ounces of absolute ethanol per day | .06 (.134) | .131 (.181) | .4 (.465)
Statistical Analysis 1: Comparison: Affective Training vs Neutral Training vs Control (Non-active); Test type: Superiority; p = .212, ANOVA

11. Secondary Outcome: Moos Health and Daily Living Scale
Description: Summarizes responses to 14 different topics that may cause disagreements in the participants' family. Response to each topic is binarized (Yes = 1; No = 0). Single summary score is generated by summing across all topics. The maximum score is 14; the minimum score is 0. Higher values represent a worse outcome.
Time Frame: 30 days following post-training assessment, up to 1.5 months
Measure: Mean (Standard Deviation); unit: units on a scale (disagreements)
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Number analyzed (Participants) | 6 | 5 | 4
units on a scale (disagreements) | 1.33 (1.03) | .4 (.548) | .25 (.5)
Statistical Analysis 1: Comparison: Affective Training vs Neutral Training vs Control (Non-active); Test type: Superiority; p < .001, ANOVA

12. Secondary Outcome: Change in Profile of Mood States
Description: Mood/affect assessment in which participants indicate whether presented words describe how they have felt during the past week on a scale from 0-4, where 0 indicates "not at all"; 1 indicates "a little"; 2 indicates "moderately"; 3 indicates "quite a bit"; and 4 indicates "extremely". The outcome reflects a difference in total score from pre- to post-test, with negative values reflecting improvements.
Time Frame: Approximately 30 days following post-training assessment, up to 1.5 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Number analyzed (Participants) | 6 | 6 | 4
score on a scale | -12.7 (37.9) | 6.67 (15.6) | 1.25 (12.3)
Statistical Analysis 1: Comparison: Affective Training vs Neutral Training vs Control (Non-active); Test type: Superiority; p = .445, ANOVA

13. Secondary Outcome: Mini Alcohol Craving Experience Questionnaire
Description: Indexes alcohol craving frequencies. Questions include:
  1. Over the past week, how often did you have a strong urge to drink?
  2. Over the past week, how often did you picture alcohol or drinking?
  3. Over the past week, how often did you imagine what it would taste like?
  4. Over the past week, how often did you imagine how your body would feel if you had a drink?
     Higher scores reflect greater craving.
  5. Over the past week, how often were these thoughts intrusive?
  Participants respond on a scale from 1-10 for each question. Responses are summed. Thus, scores range from 5-50.
Time Frame: 30 days following post-training assessment, up to 1.5 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
Number analyzed (Participants) | 6 | 6 | 5
units on a scale | 15.7 (10.7) | 10 (9.65) | 5.2 (8.98)
Statistical Analysis 1: Comparison: Affective Training vs Neutral Training vs Control (Non-active); Test type: Superiority; p = .245, ANOVA

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 weeks.
Arm/Group | Affective Training | Neutral Training | Control (Non-active)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT03137654/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT03137654/ICF_001.pdf